CLINICAL TRIAL: NCT05537519
Title: Phage Therapy for the Treatment of Urinary Tract Infection
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Applied Health Research Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Phage Therapy 001
Record Dates: First submitted 2022-09-09; First posted 2022-09-13 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Recurrent Urinary Tract Infection
Keywords: Phage Therapy; Recurrent urinary tract infection
MeSH Terms: conditions — Urinary Tract Infections | interventions — Phage Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open Label Arm (Experimental)
  Interventions: Biological: Phage Therapy

INTERVENTIONS:
Biological: Phage Therapy — 3-phage cocktail comprised of HP3, HP3.1 and ES19

SUMMARY:
This is a single-patient, phase I/II clinical trial that aims to evaluate the potential of bacteriophage therapy to treat and prevent the recurrence of a drug-resistant urinary tract infection with serious long-term effects. This study will follow a minimally invasive phage therapy approach consisting of oral, topical (opening of the urethra) and bladder installations of a 3-phage cocktail comprised of HP3, HP3.1 and ES19.

DETAILED DESCRIPTION:
This is a single-patient, phase I/II clinical trial that aims to evaluate the potential of bacteriophage therapy to treat and prevent the recurrence of a drug-resistant urinary tract infection. This study will follow a minimally invasive phage therapy approach consisting of oral, topical and bladder installations of a 3-phage cocktail comprised of HP3, HP3.1 and ES19.

Oral and bladder installation of bacteriophages will be administered on day 1 - and potentially day 7 depending on day 5 urine and stool lab results - and a topical preparation will be applied externally to the urethra for 30-minutes on days 1 to 3. However, if the participant is still experiencing mild symptoms on day 5, systemic antibiotics will be administered in combination with phage therapy.

The primary objective is to determine the safety and tolerability of minimally invasive bacteriophage therapy for treating recurrent urinary tract infections with severe long-term effects.

The secondary objective is to evaluate the 90-day clinical and microbial response to the minimally invasive administration of bacteriophages for recurrent urinary tract infections with severe long-term outcomes.

The total duration of participant involvement is 2 years, while the study is estimated to be completed in 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of recurrent chronic urinary tract infections with severe long term effects
* Can speak and understand English
* Willing to follow the protocol

Exclusion Criteria:

* Stage 5 chronic kidney disease
* Abnormal liver function tests
* A urinary stent or chronic indwelling catheterization
* A known allergy to phage products
* Fever
* Pregnancy
* Involved in another clinical trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 90 Days
  The primary objective is to determine the safety and tolerability of minimally invasive bacteriophage therapy for treating recurrent urinary tract infections with severe long-term effects.
  These will be assessed through the use of a daily symptom questionnaire, adverse events (AEs), clinical and research laboratory results.

SECONDARY OUTCOMES:
Clinical and microbial response | 90 Days
  The secondary objective is to evaluate the 90-day clinical outcomes through a daily paper questionnaire and microbial response assessed through a series of blood, urine, stool, and vaginal sample, to the minimally invasive administration of bacteriophages for recurrent urinary tract infections with severe long-term outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory German, MD PhD FRCPC, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Joseph's Health Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No